CLINICAL TRIAL: NCT02416011
Title: Smoking Cessation Self-Help for Dual Users of Tobacco Cigarettes and E-Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18127; R01DA037961-01A1 (NIH)
Record Dates: First submitted 2015-04-01; First posted 2015-04-14 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Smoking Cessation
Keywords: e-cigarette; nicotine dependence
MeSH Terms: conditions — Smoking Cessation; Vaping; Tobacco Use Disorder | interventions — Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment Only (ASSESS) (No Intervention): Participants in this condition will not receive any intervention materials. They will participate solely in the repeated assessments. Including this comparison condition controls for the effect of repeated assessments and allows for the most meaningful evaluation of the efficacy effect size as well as the cost-effectiveness of the eTARGET intervention. This condition will also be the primary source of data for the secondary surveillance aim regarding naturalistic changes in smoking and e-cigarette use over time.
- Generic Self-Help (GENERIC) (Active Comparator): This will allow us to evaluate our novel self-help intervention for e-cigarette users (our If you Vape booklets) against a matched non-targeted intervention that has demonstrated efficacy for cigarette smokers in general. Such a comparison controls for the possibility that e-cigarette users are sufficiently primed to quit smoking and that even a generic, non-targeted intervention would be effective. This possibility will be directly tested by comparing this condition against both the ASSESS and eTARGET conditions in terms of clinical outcomes and cost-effectiveness.
  Interventions: Behavioral: GENERIC
- Targeted Self-Help (eTARGET) (Experimental): Participants in this condition will receive the intervention created as the product of Study I.
  Interventions: Behavioral: eTARGET

INTERVENTIONS:
Behavioral: GENERIC — The initial Stop Smoking for Good brochure, 10 Stop Smoking for Good booklets and 9 supportive My Story pamphlets delivered over 18 months, as used in our previous cessation study.
  Other Names: self-help
  Arms: Generic Self-Help (GENERIC)
Behavioral: eTARGET — The product of Study I is expected to include the initial If You Vape brochure, a series of 10 If You Vape: Guide to Quitting Smoking booklets, distributed over 18 months, and 9 supportive My Story pamphlets, delivered in the months between booklets.
  Other Names: self-help
  Arms: Targeted Self-Help (eTARGET)

SUMMARY:
The purpose of this study is to develop and test a series of booklets designed to assist smokers of tobacco cigarettes who are also using e-cigarettes (dual users) in quitting smoking and remaining smoke-free.

DETAILED DESCRIPTION:
The first two aims of the present proposal are to adapt a validated self-help, smoking-cessation intervention to meet the needs of current dual users, and to test this new intervention in a randomized controlled trial (RCT). A third primary aim is to calculate the cost-effectiveness of the intervention. A secondary aim is to gather longitudinal data regarding the patterns of tobacco and e-cigarette use and the course of cessation of either product among dual users.

Specific Aim 1. To create a minimal smoking-cessation intervention for current dual users of tobacco cigarettes and e-cigarettes (Study I). The intervention will comprise a series of booklets and pamphlets modeled after the Forever Free booklets found to be successful at producing long-term abstinence among the general population of smokers, but adapted to the special needs, circumstances, and risk factors of dual users.

Validated methodologies used for adapting the intervention mirror those used in our prior smoking cessation studies, and reflect systematic approaches across two-phases informed by individual interviews and learner verification methodologies. The intervention will provide assistance for smoking cessation, and also encourage users to taper and eventually terminate their e-cigarette use as per traditional nicotine replacement therapy (NRT). The end product of Study I will be a series of booklets tentatively titled, "If You Vape: Guide to Quitting Smoking," available both in printed and electronic formats.

Specific Aim 2. To evaluate the efficacy of the intervention via a randomized, controlled clinical trial of current dual users (Study II). We will compare the intervention developed under Specific Aim 1 with both an assessment-only condition and a generic self-help condition comprising existing smoking cessation booklets. We hypothesize that recipients of our targeted If You Vape booklets will show higher rates of tobacco abstinence at 6, 12, 18, and 24 months after enrollment, as compared to both comparison conditions. A secondary hypothesis is that the new intervention will produce higher rates of abstinence from e-cigarettes themselves. To identify mechanism of change, we will also test several a priori moderator and mediator variables, including gender, socio-economic status, motivation to quit, nicotine dependence, e-cigarette expectancies, and magnitude of e-cigarette use (frequency, dosage).

Specific Aim 3. To calculate and compare the cost-effectiveness of the interventions. Cost- effectiveness data are vital for evaluating the real-world feasibility of an intervention. Small improvements in treatment efficacy may not be justified if they require substantially greater cost. We will compare the interventions not only on outcome efficacy, but on cost-effectiveness with respect to cost per incremental cessation and expected life-years saved.

ELIGIBILITY:
Inclusion Criteria:

* Study I - First Phase - No Longer Recruiting

  * Greater than 1 year history of daily smoking
  * 1 month or more of e-cigarette use
  * Able to speak and read English
  * (1) current dual users (of tobacco cigarettes and e-cigarettes) without interest in quitting smoking; (2) current dual users who have attempted, but not quit smoking; (3) current e-cigarette users who have successfully quit smoking; and (4) former dual users who have quit both products.
* Study I - Second Phase - No Longer Recruiting

  * Current dual users (of tobacco cigarettes and e-cigarettes)
  * Smoking at least one cigarette per day over the past year
  * Using e-cigarettes at least once per week over the past month
  * Not currently enrolled in a face-to-face smoking cessation program
  * Able to speak and read English
* Study II - No Longer Recruiting

  * Current dual users (of tobacco cigarettes and e-cigarettes)
  * Smoking at least one cigarette per week over the past year
  * Using e-cigarettes at least once per week over the past month
  * Not currently enrolled in a face-to-face smoking cessation program
  * Able to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2896 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Martinez U, Simmons VN, Sutton SK, Drobes DJ, Meltzer LR, Brandon KO, Byrne MM, Harrell PT, Eissenberg T, Bullen CR, Brandon TH. Targeted smoking cessation for dual users of combustible and electronic cigarettes: a randomised controlled trial. Lancet Public Health. 2021 Jul;6(7):e500-e509. doi: 10.1016/S2468-2667(20)30307-8. PMID 34175001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Assessment Only (ASSESS) | Generic Self-Help (GENERIC) | Targeted Self-Help (eTARGET)
Started | 575 | 1154 | 1167
Completed | 561 | 1101 | 1114
Not Completed | 14 | 53 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assessment Only (ASSESS) | Generic Self-Help (GENERIC) | Targeted Self-Help (eTARGET) | Total
Number analyzed (Participants) | 575 | 1154 | 1167 | 2896
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 69 | 76 | 175
  Between 18 and 65 years | 539 | 1073 | 1085 | 2697
  >=65 years | 6 | 12 | 6 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 435 | 424 | 1066
  Male | 368 | 719 | 743 | 1830
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 87 | 89 | 241
  Not Hispanic or Latino | 510 | 1067 | 1078 | 2655
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 27 | 11 | 53
  Asian | 5 | 9 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 3 | 8 | 7 | 18
  Black or African American | 10 | 35 | 41 | 86
  White | 513 | 1012 | 1025 | 2550
  More than one race | 27 | 57 | 64 | 148
  Unknown or Not Reported | 2 | 6 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 575 | 1154 | 1167 | 2896

OUTCOME MEASURES:

1. Primary Outcome: Rate of Smoking Abstinence
Description: Percentage rate of smoking abstinence for participants who received If You Vape booklets, compared to: A) participants in an assessment-only condition; B) participants in a generic self-help condition comprising existing smoking cessation booklets.
Time Frame: 18 months & 24 months post study enrollment
Measure: Number; unit: percentage of participants
Groups:
- ASSESS at 18 Months; ASSESS at 24 Months: Participants in this condition did not receive any intervention materials.
- GENERIC at 18 Months; GENERIC at 24 Months: This allowed investigators to evaluate their novel self-help intervention for e-cigarette users (our If you Vape booklets) against a matched non-targeted intervention that has demonstrated efficacy for cigarette smokers in general.
- eTARGET at 18 Months; eTARGET at 24 Months: Participants in this condition received the intervention the If You Vape brochure, a series of 10 If You Vape: Guide to Quitting Smoking booklets, distributed over 18 months, and 9 supportive My Story pamphlets, delivered in the months between booklets.
Arm/Group | ASSESS at 18 Months | ASSESS at 24 Months | GENERIC at 18 Months | GENERIC at 24 Months | eTARGET at 18 Months | eTARGET at 24 Months
Number analyzed (Participants) | 575 | 575 | 1154 | 1154 | 1167 | 1167
percentage of participants | 33 | 40 | 37 | 42 | 38 | 42

2. Secondary Outcome: Changes in the Use of Tobacco Products
Description: As a surveillance study, investigators will track changes in the use of both tobacco cigarettes and e-cigarettes over time for ASSESS group only
Time Frame: 18 and 24 months post study enrollment
Population: For this outcome measure, only the ASSESS group was analyzed for naturalistic changes in smoking and e-cigarette use over time.
Measure: Number; unit: percentage of participants
Groups:
- Asses Cigarette Use at 18 Months; ASSES Vaping at 18 Months: Participants in this condition did not receive any intervention
- ASSESS Cigarette Use at 24 Months; ASSESS Vaping at 24 Months: Participants in this condition did not receive any intervention materials.
Arm/Group | Asses Cigarette Use at 18 Months | ASSESS Cigarette Use at 24 Months | ASSES Vaping at 18 Months | ASSESS Vaping at 24 Months
Number analyzed (Participants) | 575 | 575 | 575 | 575
percentage of participants | 33 | 40 | 27 | 32

3. Other Pre Specified Outcome: Study 2: Cost Effectiveness
Description: Cost per incremental cessation will be measured using USD spent on the self help materials provided to the participants in the Generic and eTarget groups at 18 months and 24 months. ***Total cost was calculated for the intervention and not calculated as per participant cost
Time Frame: 18 months and 24 months after study recruitment
Population: Participant groups evaluated at 18 and 24 months
Measure: Number; unit: USD
Groups:
- ASSESS Group at 18 Months: Participants in this condition did not receive any intervention materials
- ASSESS Group at 24 Months: Participants in this condition did not receive any intervention
- GENERIC Group at 18 Months; GENERIC Group at 24 Months: This group allowed investigators to evaluate their novel self-help intervention for e-cigarette users (If you Vape booklets) against a matched non-targeted intervention that has demonstrated efficacy for cigarette smokers in general.
- eTARGET Group at 18 Months; eTarget Group at 24 Months: Participants in this condition received the intervention; If You Vape brochure, a series of 10 If You Vape: Guide to Quitting Smoking booklets, distributed over 18 months, and 9 supportive My Story pamphlets, delivered in the months between booklets.
Arm/Group | ASSESS Group at 18 Months | ASSESS Group at 24 Months | GENERIC Group at 18 Months | GENERIC Group at 24 Months | eTARGET Group at 18 Months | eTarget Group at 24 Months
Number analyzed (Participants) | 575 | 575 | 1154 | 1154 | 1167 | 1167
USD | 0 | 0 | 1535 | 2369 | 1000 | 2253

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected
Description: Participants were not given any type of drug. The intervention participants received was the If You Vape brochure, a series of 10 If You Vape: Guide to Quitting Smoking booklets and 9 supportive My Story pamphlets
Arm/Group | Assessment Only (ASSESS) | Generic Self-Help (GENERIC) | Targeted Self-Help (eTARGET)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02416011/Prot_SAP_000.pdf